CLINICAL TRIAL: NCT01933009
Title: The Effect of GnRH Administration During Luteal Support in Frozen-thawed Transfer Cycles
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Dr. Ido Ben-Ami, MD PhD, Assaf-Harofeh Medical Center
Other Study IDs: 79/13
Record Dates: First submitted 2013-08-28; First posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Pregnancy Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

SUMMARY:
GnRH administration during the luteal phase was found to significantly increase pregnancy rates in women undergoing fresh-cycle IVF cycles.

We aim to investigate the effect of GnRH administration during the luteal phase in women undergoing frozen-thawed IVF cycles.

ELIGIBILITY:
Inclusion Criteria:

Frozen-thawed IVF cycles

Exclusion Criteria:

Hydrosalpings Uterine myomas

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women undergoing frozen-thawed IVF cycles
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-05 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- IVF and infertility unit, Assaf Harofeh Medical Center, Ẕerifin, Be'er-Ya'akov, Israel